CLINICAL TRIAL: NCT00881309
Title: To Compare the Efficacy and Safety of Tripterygium (TW) vs Aza in the Maintenance Therapy for Lupus Nephritis
Brief Title: To Compare the Efficacy and Safety of Tripterygium (TW) Versus AZA in the Maintenance Therapy for Lupus Nephritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Weixin Hu, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0902
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2009-04

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- immunosuppressor (Experimental)
  Interventions: Drug: Tripterygium

INTERVENTIONS:
Drug: Tripterygium — TW 90mg/d

SUMMARY:
The purpose of this study is to:

* To access the efficacy of TW compared to Aza in the maintenance therapy for lupus nephritis
* To investigate the safety and tolerability of TW versus Aza in the maintenance therapy for lupus nephritis

DETAILED DESCRIPTION:
Tripterygium (TW) is a Chinese traditional patent drugs in treating chronic glomerulonephritis. It has been used to treat lupus nephritis for many years with less side effects. We compare the efficacy and safety of TW vs Aza in the maintenance therapy of lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who signed written informed consent form;
2. SLE patient, aged between 18-60 years, female or male;
3. Patients diagnosed lupus nephritis according to ISN/RPS 2003 classification criteria, class Ⅲ, Ⅳ,Ⅳ+Ⅴ, Ⅲ+Ⅴ or Ⅴ LN by renal biopsy;
4. All patients received induction therapy for 6-12 months, including MMF, CTX, FK506 or multi-target therapy;
5. When recruited in the study, patients received partial remission or complete remission for 3 months;

   * Complete remission: proteinuria < 0.4 g/24h, negative urine sediment, serum albumin > 35 g/L, elevated scr < 0.3 mg/dl, no extra-renal complications;
   * Partial remission: proteinuria < 1.0 g/24h, urine RBC < 500000/ml without casts, serum albumin > 35 g/L, elevated scr <0.3 mg/dl, no extra-renal complications.

Exclusion Criteria:

1. Patients who didn't sign written informed consent form or could not obey the protocol;
2. Patients who didn't received the CR or PR criterion;
3. Patients who have impaired liver function, with ALT/GPT or AST/GOT twice more than the normal upper limit;
4. WBC < 3000/mm3 in peripheral blood;
5. Patients with abnormal of central nervous system.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
complete remission rate | 2 years

SECONDARY OUTCOMES:
renal relapse | 2 years
partial remission | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Weixin Hu, Doctor, Principal Investigator — Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology,Jinling Hospital, Nanjing, Jiangsu, China